CLINICAL TRIAL: NCT02990559
Title: Neuroimaging of Donor Iron Deficient Study (DIDS)
Brief Title: Neuroimaging of Donor Iron Deficient Study
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Eldad Arie Hod, Associate Professor of Pathology and Cell Biology, Dept of Pathology&Cell Biology, Columbia University
Other Study IDs: AAAR0145
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Iron Deficiency
Keywords: Iron repletion; Blood donation; Transfusion
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Iron Repletion: Subjects participating in the associated study under the Iron Repletion arm will also undergo MRI (Magnetic Resonance Imaging) scan/fMRI (functional Magnetic Resonance Imaging) scan on two occasions, while performing cognitive tasks.
- Placebo: Subjects participating in the associated study under the Placebo arm will also undergo MRI/fMRI scans on two occasions, while performing cognitive tasks.

SUMMARY:
This pilot study is designed to investigate (1) whether getting iron treatment affects iron in the brain and (2) how getting iron treatment affects brain functions when it is performing specific cognitive tasks. By cognitive tasks, it means tasks that involve perceiving, representing, or assessing things. The specific cognitive tasks used here will involve tests of memory and processing speed.

DETAILED DESCRIPTION:
Iron, the most abundant metal in the brain, is vital for multiple cellular processes, including neurotransmitter synthesis, neuron myelination, and mitochondrial function. In the United States, of the donors who provided the ~15 million units of red blood cells that were collected for transfusion, 69% were repeat donors. Although iron deficiency is surprisingly prevalent in first-time donors, its prevalence is even higher in these particularly altruistic frequent donors, (i.e., up to 49% and 66% of male and female repeat donors, respectively), manifested as iron depletion or iron-deficient erythropoiesis. Iron deficiency from blood donation is associated with fatigue, restless leg syndrome, decreased physical endurance and work capacity, and impaired concentration, attention, and other neurocognitive functions; however, these conclusions are not based on definitive studies and have not yet changed blood donation policy. This study is to collect data through noninvasive procedures routinely employed in clinical practice to better understand how iron treatment may affect brain functions.

ELIGIBILITY:
Inclusion Criteria:

* Current participant of the associated randomized controlled trial conducted at Columbia University Medical Center (therefore invited to participate in this optional ancillary study).

Exclusion Criteria:

* Not a current participant of the associated randomized controlled trial conducted at Columbia University Medical Center.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with iron deficiency from blood donation will be recruited over 5 years in the associated randomized controlled trial conducted at Columbia University Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Change in mean iron content in specific brain nuclei | Up to 5 months
  To assess the iron deposition/accumulation in subjects' brain region by using neuroimaging such as MRI/fMRI.
Cognition Fluid Composite Score | Up to 5 months
  NIH Toolbox derived uncorrected standard composite score, measured at 4 time points (twice pre-randomization and twice post-randomization). The uncorrected standard score will be used, where the normative mean is 100 with a standard deviation of 15.

SECONDARY OUTCOMES:
Activity and connectivity in specific functional networks at resting state | Up to 5 months
  Resting state blood oxygen level dependent (BOLD) signals will be assessed by fMRI. Independent component analysis will be used to detect alterations in connectivity in functional networks (e.g., default mode network and visual, sensory/motor, executive control, temporal/parietal, basal ganglia components) in a paired analysis comparing subjects before and after iron repletion versus placebo.
Brain activity during tasks of processing speed and episodic memory | Up to 5 months
  Brain activity patterns during performance of processing speed and episodic memory tasks will be assessed by fMRI and comparisons made from before to after iron repletion versus placebo.
NIH Toolbox Auditory Verbal Learning Test (Rey) Score | Up to 5 months
  NIH Toolbox derived uncorrected standard Auditory Verbal Learning test score, measured at 4 time points (twice pre-randomization and twice post-randomization). Delayed and initial scores analyzed separately. The raw score will be used in which a higher number represents more words remembered.
NIH Toolbox Flanker Inhibitory Control and Attention Test Score | Up to 5 months
  NIH Toolbox derived uncorrected standard Flanker Inhibitory Control and Attention test score (single score), measured at 4 time points (twice pre-randomization and twice post-randomization). The uncorrected standard score will be used, where the normative mean is 100 with a standard deviation of 15.
NIH Toolbox List Sorting Working Memory Test Score | Up to 5 months
  NIH Toolbox derived uncorrected standard List Sorting Working Memory test score, measured at 4 time points (twice pre-randomization and twice post-randomization). The uncorrected standard score will be used, where the normative mean is 100 with a standard deviation of 15.
NIH Toolbox Dimensional Change Card Sort Test | Up to 5 months
  NIH Toolbox derived uncorrected standard Dimensional Change Card Sort test score, measured at 4 time points (twice pre-randomization and twice post-randomization). The uncorrected standard score will be used, where the normative mean is 100 with a standard deviation of 15.
NIH Toolbox Pattern Comparison Processing Speed Test Score | Up to 5 months
  NIH Toolbox derived uncorrected standard Pattern Comparison Processing Speed test score, measured at 4 time points (twice pre-randomization and twice post-randomization). The uncorrected standard score will be used, where the normative mean is 100 with a standard deviation of 15.
NIH Toolbox Picture Sequence Memory Test | Up to 5 months
  NIH Toolbox derived uncorrected standard Picture Sequence Memory test score, measured at 4 time points (twice pre-randomization and twice post-randomization). The uncorrected standard score will be used, where the normative mean is 100 with a standard deviation of 15.

CONTACTS AND LOCATIONS:
Overall Officials: Eldad Hod, MD, Principal Investigator — Associate Professor of Pathology and Cell Biology, Dept of Pathology&Cell Biology
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hare D, Ayton S, Bush A, Lei P. A delicate balance: Iron metabolism and diseases of the brain. Front Aging Neurosci. 2013 Jul 18;5:34. doi: 10.3389/fnagi.2013.00034. eCollection 2013. PMID 23874300
- [Background] Smith GA, Fisher SA, Doree C, Roberts DJ. A systematic review of factors associated with the deferral of donors failing to meet low haemoglobin thresholds. Transfus Med. 2013 Oct;23(5):309-20. doi: 10.1111/tme.12046. Epub 2013 Jul 5. PMID 23829880
- [Background] Bialkowski W, Bryant BJ, Schlumpf KS, Wright DJ, Birch R, Kiss JE, D'Andrea P, Cable RG, Spencer BR, Vij V, Mast AE. The strategies to reduce iron deficiency in blood donors randomized trial: design, enrolment and early retention. Vox Sang. 2015 Feb;108(2):178-85. doi: 10.1111/vox.12210. Epub 2014 Dec 3. PMID 25469720
- [Background] Cable RG, Glynn SA, Kiss JE, Mast AE, Steele WR, Murphy EL, Wright DJ, Sacher RA, Gottschall JL, Tobler LH, Simon TL; NHLBI Retrovirus Epidemiology Donor Study-II (REDS-II). Iron deficiency in blood donors: the REDS-II Donor Iron Status Evaluation (RISE) study. Transfusion. 2012 Apr;52(4):702-11. doi: 10.1111/j.1537-2995.2011.03401.x. Epub 2011 Oct 24. PMID 22023513
- [Background] Brittenham GM. Iron deficiency in whole blood donors. Transfusion. 2011 Mar;51(3):458-61. doi: 10.1111/j.1537-2995.2011.03062.x. No abstract available. PMID 21388389
- [Background] Newman B. Iron depletion by whole-blood donation harms menstruating females: the current whole-blood-collection paradigm needs to be changed. Transfusion. 2006 Oct;46(10):1667-81. doi: 10.1111/j.1537-2995.2006.00969.x. No abstract available. PMID 17002622
- [Derived] Hod EA, Habeck C, Zhuang H, Dimov A, Spincemaille P, Kessler D, Bitan ZC, Feit Y, Fliginger D, Stone EF, Roh D, Eisler L, Dashnaw S, Caccappolo E, McMahon DJ, Stern Y, Wang Y, Spitalnik SL, Brittenham GM. Effects of iron repletion on brain iron content, myelination, neural network activation, and cognition. JCI Insight. 2025 Oct 21;10(23):e194442. doi: 10.1172/jci.insight.194442. eCollection 2025 Dec 8. PMID 41118254
- [Derived] Hod EA, Brittenham GM, Bitan ZC, Feit Y, Gaelen JI, La Carpia F, Sandoval LA, Zhou AT, Soffing M, Mintz A, Schwartz J, Eng C, Scotto M, Caccappolo E, Habeck C, Stern Y, McMahon DJ, Kessler DA, Shaz BH, Francis RO, Spitalnik SL. A randomized trial of blood donor iron repletion on red cell quality for transfusion and donor cognition and well-being. Blood. 2022 Dec 22;140(25):2730-2739. doi: 10.1182/blood.2022017288. PMID 36069596